CLINICAL TRIAL: NCT00499187
Title: A Preliminary Evaluation of Fanconi Syndrome Due to Antiretroviral Therapies in HIV-Infected Persons
Brief Title: Fanconi Syndrome Due to ARVs in HIV-Infected Persons
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-104-0353
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections; Fanconi Syndrome; Kidney Disease; Renal Impairment
Keywords: Fanconi; Kidney; Renal; HIV; HIV-1; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Fanconi Syndrome; Kidney Diseases; Renal Insufficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fanconi Cases: This cohort enrolled participants with evidence of protocol-defined Fanconi syndrome (confirmed creatinine clearance decline and evidence of proximal tubulopathy).
  Interventions: Procedure: Blood Draws
- Control Cases: This cohort enrolled participants with no evidence of protocol-defined Fanconi syndrome.
  Interventions: Procedure: Blood Draws

INTERVENTIONS:
Procedure: Blood Draws — A single whole blood sample was collected for genomic analysis.

SUMMARY:
Cross-sectional cohort study of participants with HIV with or without protocol-defined Fanconi syndrome (confirmed creatinine clearance [CLcr] decline and evidence of proximal tubulopathy).

ELIGIBILITY:
Inclusion Criteria - Fanconi Cases

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

* Adult (greater than or equal to 18 years) HIV-1 infected subjects regardless of race or ethnicity.
* Subjects must be on a stable ARV regimen for greater than or equal to 1 month prior to study entry.
* Evidence of protocol-defined Fanconi syndrome
* TDF subjects must be on TDF-containing regimen at the time of onset of Fanconi syndrome.
* Negative serum pregnancy test (females of child-bearing potential only).
* Less than two years post-menopausal women of child-bearing potential (TDF subjects only) agree to follow an adequate birth control barrier method or agree to abstain from heterosexual intercourse while participating in the study.
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Exclusion Criteria - Fanconi Cases

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

* Non TDF subjects who have received any TDF within the prior 6 months, or those who have received greater than 2 weeks cumulative treatment.
* TDF subjects who have previously served as a TDF control for this protocol.
* History of current alcohol or substance abuse judged by the investigator to potentially interfere with laboratory results.

Inclusion Criteria - Controls

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

* Adult (greater than or equal to 18 years) HIV-1 infected subjects regardless of race or ethnicity.
* No evidence of protocol-defined Fanconi syndrome
* On a TDF-containing regimen matched to a Fanconi case by clinic location, duration on TDF and age.
* Negative serum pregnancy test (females of child-bearing potential only).
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Exclusion Criteria - Controls

Subjects who meet the following exclusion criteria are not to be enrolled in this study.

• History of current alcohol or substance abuse judged by the investigator to potentially interfere with laboratory results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected subjects with protocol defined Fanconi Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Time to TDF discontinuation after diagnosis of Fanconi syndrome | Up to 48 weeks
Time to confirmed resolution of Fanconi syndrome | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (13):
- United States (10):
  - Los Angeles, California
  - Denver, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - University of Indiana, Indianapolis, Indiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - New York, New York
  - Cleveland, Ohio
  - Houston, Texas
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec